CLINICAL TRIAL: NCT06080386
Title: UDFF Performance Evaluation ((Ultrason Derived Fat Fraction)
Acronym: UDFF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: 202300122
Record Dates: First submitted 2023-10-06; First posted 2023-10-12 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Non Alcoholic Fatty Liver Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- one group: Patients who had during their care UDFF ultrasound measurements and liver MRI over the study period may be included in this study
  Interventions: Diagnostic Test: UDFF

INTERVENTIONS:
Diagnostic Test: UDFF — quantification of liver fat: UDFF (lipid fraction derived from ultrasound) from one of the probes of an ultrasound system

SUMMARY:
The purpose of this study is to assess UDFF performance (compared to MRI)

ELIGIBILITY:
Inclusion Criteria:

* All patients who had hepatic ultrasound with available UDFF measurements and hepatic MRI (with steatosis quantification sequences) between 01/01/2022 and 31/09/2023 may be included.

Exclusion Criteria:

* chronic liver disease with a different etiology other than NAFL/NASH or mixed (hepatitis B or C, hemochromatosis, autoimmune hepatitis, Wilson's disease, cholestasic disease, alpha 1 antitrypsin deficiency),
* decompensated cirrhosis (ascites, jaundice, encephalopathy, rupture of esophageal varices),
* hepatocellular carcinoma.
* opposition to the use of its data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients followed by the department of hepato gastroenterology of the CHU d'Angers for liver disease (NAFLD)
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-10-15 (Estimated)

PRIMARY OUTCOMES:
To evaluate the perfomances of the UDFF system for the quantification of hepatic steatosis in patients suspected of chronic hepatophyte. | 3 months maximum between the 2 measurements (UDFF and MRi)
  Steatosis value measured by multiecho sequences in MR

CONTACTS AND LOCATIONS:
Locations (1):
- Angers university hospital, Angers, France

IPD SHARING:
Plan to Share IPD: No